CLINICAL TRIAL: NCT05726396
Title: A Pilot Study Testing the Safety and Feasibility of Restorative Microbiota Therapy (RMT) in Patients With Refractory Immune-checkpoint Inhibitor-related Colitis
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: MNCCTN025
Record Dates: First submitted 2023-02-04; First posted 2023-02-13 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Immune-related Colitis; Colitis
MeSH Terms: conditions — Colitis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- RMT group (Experimental): 16 patients will be randomized to Oral restorative microbiota therapy (RMT). Consenting eligible participants receive a loading dose of RMT capsules.
  Interventions: Drug: RMT
- active placebo (Placebo Comparator): participants in the placebo arm will receive an identical looking placebo capsules
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: RMT — A single loading dose of RMT capsules containing ~5 x 10 11 bacteria on day 1 followed by 2 x 10 11 bacteria daily for 6 days. The RMT capsule preparation (~2-5 capsules, size 00) is self-administered on an empty stomach with at least one glass of water. Clear liquids are allowed, and food can be resumed 2 hours after administration.
  Arms: RMT group
Drug: Placebo — Participants will receive an identical looking placebo capsules daily for 7 days (i.e 5 placebo capsules on day 1), followed by 2 placebo capsules daily from Day 2-7. The placebo capsule preparation is self-administered on an empty stomach with at least one glass of water. Clear liquids are allowed, and food can be resumed 2 hours after administration.
  Arms: active placebo

SUMMARY:
Immune-related colitis from immune checkpoint inhibitors (ICI) is a common adverse effect causing significant morbidity and impairment of quality of life (QoL). Steroids are the first line of treatment for severe ICI induced Immune- mediated diarrhea and colitis (IMDC). If there is no improvement in 48 to 72 hours, other immunosuppressive agents (infliximab, vedolizumab) are recommended. However, efficacy data supporting the use of immunosuppressives for steroid refractory IMDC is limited by case reports/series. Clinical trials focusing on steroid-refractory colitis are sparse. Novel treatments for IMDC outside of blanket immunosuppression are needed. There is robust evidence to suggest that gut microbial diversity and composition is associated with both ICI efficacy and toxicity. Preliminary studies have shown that pathophysiology of immune mediated colitis may be related to loss of gut microbial diversity. Recently, multiple case series have shown the utility of fecal microbiota transplant for treatment of refractory IMDC providing the proof of concept. This is a pilot randomized placebo controlled study to assess the safety and feasibility of oral restorative microbiota therapy (RMT) in patients with steroid- refractory IMDC.

ELIGIBILITY:
Inclusion Criteria:

* Localized, locally advanced or metastatic solid tumors who have received at least two doses of ICI (PD-1/PD-L1 with or without CTLA-4 inhibitor).
* ICI used as a single agent, or combination or ICI in combination with other cytotoxic chemotherapy or targeted therapy for curative or palliative intent treatment.
* Last ICI treatment with in 6 weeks of onset of IMDC symptoms
* Meet one of the criteria for steroid refractory IMDC defined as:

  1. Persistent symptoms (NCI CTCAE v 5.0 Grade ≥ 2 diarrhea) following high-dose corticosteroid therapy (≥1 mg/kg/day prednisone or equivalent) for least 48 hours or
  2. Persistent symptoms (ongoing Grade ≥ 2 diarrhea per CTCAE v5.0.) following use of a one or more biologic agent (i.e. either a TNFα inhibitor or an anti-integrin) in addition to corticosteroids (with starting dose of prednisone or equivalent ≥1 mg/kg/day for at least 48 hours followed by receipt of at least one dose of either a TNFα inhibitor or an anti- integrin for at least 48 hours or
  3. For patients with relapsed IMDC who have discontinued steroids: Relapsed IMDC symptoms for 24 or more hours (NCI CTCAE v 5.0 Grade ≥ 2 diarrhea) within 4 weeks of discontinuing prednisone or equivalent. These patients should have received initial high-dose corticosteroid therapy (˃1 mg/kg/day prednisone or equivalent) with subsequent taper over at least 4 weeks or
  4. For patients with relapsed IMDC following the tapering of steroids Relapsed IMDC symptoms for 24 or more hours (NCI CTCAE v 5.0 Grade ≥ 2 diarrhea) while the prednisone taper is on-going. These patients should have received initial high-dose corticosteroid therapy (˃1 mg/kg/day prednisone or equivalent) with resulting clinical resolution of diarrhea (NCI CTCAE v 5.0 Grade ˂ 1 diarrhea) for at least 24 hours before relapse
* Adequate organ function within 14 days prior to study enrollment defined as:

  1. Hematology: Hemoglobin ≥9.0 g/dL, absolute neutrophil count (ANC) ≥1,000/mcL, platelets ≥75,000/mcL,
  2. Hepatic function: Total bilirubin ≤ 1.5x upper limit of normal (ULN), AST (SGOT) and ALT (SGPT) ≤ 2.5 x institutional ULN unless liver metastases are present, in which case it must be ≤5x ULN)
  3. Renal function: measured creatinine clearance >40 mL/min or estimated glomerular filtration rate (GFR) >40 mL/min If AST/ALT and serum creatinine elevation are suspected to be irAEs, patients are eligible as long as the irAE are controlled (i.e. not getting worse at the time of enrollment)
* Well controlled diabetes with HbA1c of <8 with in 6 months of screening
* Euvolemic on physical examination
* Stable vital signs at screening and enrollment that includes

  1. Body temperature 95.8 to 99.9°F
  2. Heart rate between 60-100/min
  3. Blood pressure 90-140/60-90 mm of Hg.
* Must be on standard antidiarrheal supportive care for at least 1 day prior to starting RMT. The regimen consists of: loperamide 2-4 mg every 6 hours (up to 16 mg /day) and/or diphenoxylate 5 mg/ atropine sulfate 0.05 mg (2 tabs or 10 ml) up to 4 times daily as needed. This will continue until resolution of diarrhea to NCI CTCAE v 5.0 Grade ≤ 1.
* Age 18 years of age or older at the time of consent
* Body weight of >30 kg
* Expected survival for at least 6 months in the opinion of the enrolling investigator as documented in the medical record
* Voluntary written consent prior to the performance of any research related activity.

Exclusion Criteria:

* Diagnosis of concomitant infectious colitis based on standard stool screening including stool microscopy for ova and parasites, stool PCR for Clostridioides difficile, and locally available common enteric bacterial pathogen and viral panel by PCR.
* Last cytotoxic chemotherapy or targeted therapy less than 3 week prior to screening
* Patients anticipated to require cytotoxic chemotherapy or targeted therapy through the end of treatment EOT period (30 days following first dose of RMT)
* Known current pregnancy or breastfeeding.
* Receiving another investigational agent or has received an investigational agent within 60 days of study enrollment.
* Any other uncontrolled Grade ≥3 infection at the time of enrollment (Concomitant systemic antibiotics for non-GI infections are allowed).
* Previous documented history of chronic diarrhea from non-IMDC causes (For example: inflammatory bowel disease (e.g., Crohn's disease, ulcerative colitis).
* Known dysphagia or inability to swallow study capsules (CTCAE v5 Dysphagia Grade ≥2 - symptomatic and altered eating/swallowing).
* Known risk of aspiration based on history or current complaints.
* Has a known sensitivity to any component of therapeutic agents used in this study.
* On intravenous biologic agents for other baseline autoimmune conditions.
* Other concomitant uncontrolled irAE's at the time of enrollment which would require systemic corticosteroids or biologic immunomodulatory agents.
* On chronic systemic antibiotic therapy (antibiotics for ≥60 consecutive days within 12 weeks of enrollment).
* Receipt of over-the-counter probiotics in the last 4 weeks
* Receipt of live attenuated vaccination within 30 days of receiving RMT. Examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, chickenpox (except shingrix), yellow fever, nasal seasonal flu, nasal H1N1 flu, rabies, BCG, and typhoid - COVID-19 vaccination is permitted.
* Psychiatric illness/social situations that would limit compliance with study requirements or compromise the ability of the patient to give written informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-09-23 (Actual); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
Feasibility and safety of RMT | 6 months after baseline
  Feasibility and safety of RMT as assessed by the occurrence of adverse events

SECONDARY OUTCOMES:
Clinical remission by Day 10 | Day 10
  Proportion of patients who experience diarrhea resolution to Grade <= 1 of refractory IMDC at Day 10 from 1st dose of RMT
Clinical remission by Day 30 | Day 30
  Incidence of clinical remission of refractory IMDC at Day 30 following first dose of RMT
Time for clinical remission | Day 180
  Days to induce a clinical remission of refractory IMDC necessary to achieve a diarrhea of Grade <= 1

CONTACTS AND LOCATIONS:
Overall Officials: Ajay Prakash, MD, PhD, Principal Investigator — University of Minnesota
Locations (9):
- United States (9):
  - Essentia Health St. Joseph's Medical Center, Brainerd, Minnesota
  - Essentia Health Deer River Clinic, Deer River, Minnesota
  - Essentia Health St. Mary's Detroit Lakes Clinic, Detroit Lakes, Minnesota
  - Essentia Health Cancer Center, Duluth, Minnesota
  - Essentia Health Fosston, Fosston, Minnesota
  - Essentia Health Hibbing Clinic, Hibbing, Minnesota
  - University of Minnesota, Minneapolis, Minnesota
  - Essentia Health Sandstone, Sandstone, Minnesota
  - Essentia Health Virginia Clinic, Virginia, Minnesota